CLINICAL TRIAL: NCT05412017
Title: EPIC: Evaluation of Pharmacy-based Identification and Treatment of HCV
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cool Aid Community Health Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IN-CA-987-5735
Record Dates: First submitted 2022-05-03; First posted 2022-06-09 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C
Keywords: hepatitis C; Pharmacy; Testing
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hepatitis C Point of Care Testing and Treatment — Pharmacy led hepatitis C point of care testing

SUMMARY:
The research project aims to understand how pharmacies can be involved in the identification and treatment of hepatitis C (hep C). The study will look at the effectiveness of hep C testing and treatment through pharmacies with support from the Cool Aid Community Health Centre (CACHC). The study will also evaluate the readiness of pharmacies to take on these extra tasks at the pharmacy. This information will be used to develop future strategies to better detect, treat and prevent hep C.

DETAILED DESCRIPTION:
The primary objective of this project is to decrease barriers to care for hepatitis C (HCV) treatment for people who use drugs through the use of rapid diagnostic testing technologies, and task shifting HCV testing and treatment follow up to include trained pharmacy staff. Secondary objectives are to evaluate interest, readiness, and effectiveness of community-based pharmacies as a location for the screening and treatment of HCV.

A prospective, longitudinal interventional cohort design will be used to enrol people who access community-based pharmacies and have tested for HCV RNA. Persons with untreated chronic HCV infection will receive direct acting antiviral treatment. This is a trial of pharmacist-led HCV testing and treatment versus conventional care in HCV positive patients.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Age > 18 years old
3. Documented HCV RNA test, interested in being tested for HCV antibody or at risk for HCV (ie. "Baby boomers": anyone born between 1945-1965, anyone known to currently (past 6 months) or have a history of injecting drugs, including anyone receiving Opiate Agonist Therapy (OAT), any gay or bisexual men who have sex with men (gbMSM))

Exclusion Criteria:

1) Declined to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
HCV access to care for HCV testing and treatment | 24 weeks
  Number of patients tested for hepatitis C (HCV) antibodies through through the use of rapid diagnostic testing technologies by trained pharmacy staff that are found positive for HCV RNA and treated for HCV

CONTACTS AND LOCATIONS:
Overall Officials: Chris Fraser, MD, Principal Investigator — Medical Director
Locations (1):
- Cool Aid Community Health Centre, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No